CLINICAL TRIAL: NCT07056842
Title: A Single-Center, Open-Label, Single-Arm, Fixed-Sequence Phase I Clinical Study to Evaluate the Effect of Multiple Doses of Rifampin or Itraconazole on the Pharmacokinetics of VCT220 in Healthy Subjects
Brief Title: This is an Open-label, Non-randomized Study to Assess the Pharmacokinetics (PK) of VCT220 in Healthy Volunteers When Administered With Rifampin or Itraconazole
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vincentage Pharma Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VCT220-I-04-02
Record Dates: First submitted 2025-06-29; First posted 2025-07-09 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Obesity &Amp; Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — Rifampin; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental)
  Interventions: Drug: Rifampin + VCT220; Drug: Itraconazole + VCT220

INTERVENTIONS:
Drug: Rifampin + VCT220 — Participants will receive a single oral dose of VCT220 160 mg on Day 1. Rifampin 600 mg will be administered once daily from Day 4 to Day 10 and from Day 12 to Day 14. On Day 11, rifampin 600 mg will be administered followed 30 minutes later by VCT220 160 mg. All doses are administered under fed or fasting conditions with standardized restrictions on fluid and food intake.
Drug: Itraconazole + VCT220 — Participants will receive a single oral dose of VCT220 40 mg on Day 1. Itraconazole 200 mg will be administered once daily from Day 4 to Day 11 and from Day 13 to Day 14. On Day 12, VCT220 40 mg will be co-administered with itraconazole 200 mg after breakfast. All doses are administered under fed conditions with standardized fluid and fasting controls.

SUMMARY:
This is a single-center, open-label, single-arm, fixed-sequence Phase I study in healthy participants to evaluate the effect of multiple doses of rifampin or itraconazole on the pharmacokinetics (PK) of VCT220 and its metabolite VCT289. Cohort 1 will assess the impact of rifampin (600 mg once daily) on VCT220 (160 mg single dose). Cohort 2 will assess the impact of itraconazole (200 mg once daily) on VCT220 (40 mg single dose). A total of 32 healthy subjects will be enrolled, 16 in each cohort.

DETAILED DESCRIPTION:
This is a single-center, open-label, single-arm, fixed-sequence Phase I clinical study designed to evaluate the effect of multiple doses of rifampin or itraconazole on the pharmacokinetics (PK) of VCT220 and its primary metabolite, VCT289, in healthy subjects. The study includes two cohorts.

Cohort 1 (Rifampin group):

Participants will receive a single oral dose of VCT220 160 mg on Day 1. Rifampin 600 mg will be administered once daily from Day 4 to Day 10 and from Day 12 to Day 14. On Day 11, participants will receive rifampin 600 mg followed 30 minutes after breakfast by VCT220 160 mg. All doses will be administered under fed or fasting conditions as specified, with restrictions on fluid intake and fasting periods post-dose to standardize absorption conditions.

Cohort 2 (Itraconazole group):

Participants will receive a single oral dose of VCT220 40 mg on Day 1. Itraconazole 200 mg will be administered once daily from Day 4 to Day 11 and from Day 13 to Day 14. On Day 12, a single dose of VCT220 40 mg will be co-administered with itraconazole 200 mg after breakfast, under standardized fed conditions.

A total of 32 healthy adult subjects will be enrolled, with 16 subjects per cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Participants are able to communicate well with the investigators, fully understand the purpose, content, procedures, and potential adverse events of the study, comprehend and comply with all study requirements, and voluntarily sign the informed consent form (ICF).
2. Healthy male and female participants aged between 18 and 50 years (inclusive).
3. Male participants must weigh ≥50.0 kg, and female participants must weigh ≥45.0 kg. Body Mass Index (BMI) must be within the range of 19.0 to 28.0 kg/m² (inclusive), calculated as weight (kg)/height² (m²).
4. Participants must have no plans for conception and must voluntarily use effective contraception from the time of signing the ICF until 3 months after the last dose of study medication. No plans for sperm or egg donation during this period.

Exclusion Criteria:

1. Any clinically significant abnormalities as determined by the investigator in physical examination, vital signs, laboratory tests, abdominal ultrasound, or chest X-ray (frontal and lateral views) during screening.
2. Positive test results for HBsAg, HCV-Ab, HIV-Ab, or TPPA.
3. QTcF ≥450 ms for males or ≥470 ms for females on 12-lead ECG at screening (QTcF calculated using Fridericia's formula: QTcF = QT / RR^0.33), or clinically significant ECG abnormalities as assessed by the investigator.
4. Known allergy to VCT220, rifampin, or itraconazole, or history of hypersensitivity to two or more drugs or foods.
5. History or presence of significant diseases of the nervous, cardiovascular (unless deemed acceptable by the investigator), hematologic, lymphatic, immune, digestive, urinary, respiratory, metabolic, or musculoskeletal systems.
6. History or presence of pancreatitis (chronic or acute) or acute gallbladder disease (except those post-cholecystectomy).
7. Prior diagnosis of type 1, type 2, or other specific types of diabetes.
8. Use of GLP-1 receptor agonists within 6 months prior to screening.
9. Difficulty swallowing or any gastrointestinal disease affecting drug absorption (e.g., diarrhea, vomiting, inflammatory bowel disease, acute gastroenteritis, peptic ulcer, or chronic GI dysfunction with marked malabsorption).
10. Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2.
11. History of significant active or unstable major depression or other major psychiatric disorders within 2 years prior to screening.
12. Underwent surgery within 3 months prior to screening, plans to undergo surgery during the study period, or had surgery affecting absorption, distribution, metabolism, or excretion of drugs.
13. Participation in another drug/device clinical trial within 3 months prior to screening or planned participation during the study period.
14. Blood donation (including components) or significant blood loss ≥400 mL, receipt of blood transfusion or blood products within 3 months prior to screening.
15. Use of any prescription drugs (especially CYP3A4, CYP2C8, CYP2C9, and CYP2C19 inducers/inhibitors), over-the-counter medications, dietary supplements, or traditional Chinese medicine within 14 days prior to first dosing, or planning to use such substances during the study (excluding study medication).
16. Vaccination within 14 days prior to screening or planned vaccination during the study.
17. History of drug abuse or use of illicit drugs within 1 year prior to screening, or positive urine drug screening.
18. Smoking more than 5 cigarettes per day within 3 months prior to screening or inability to abstain from tobacco during the study.
19. Alcohol consumption >14 units/week within 3 months prior to screening (1 unit ≈ 360 mL beer at 5% alcohol, 45 mL spirits at 40%, or 150 mL wine at 12%), or inability to abstain from alcohol, or positive alcohol breath test (>0 mg/100 mL).
20. Excessive consumption of tea, coffee, or caffeinated beverages (>8 cups/day, 1 cup = 250 mL) within 3 months prior to screening, ingestion of caffeine-containing products within 24 hours before dosing, or unwillingness to abstain from caffeine during the study.
21. Consumption of fruits or products that may affect drug metabolism (e.g., pitaya, mango, grapefruit, pomelo, oranges) within 2 days prior to first dosing, or unwillingness to abstain from these during the study.
22. Special dietary requirements incompatible with standardized study meals.
23. Poor venous access or history of syncope during venipuncture or blood collection.
24. Pregnant or breastfeeding females; positive pregnancy test; or history of unprotected sex within 30 days prior to screening.
25. Use of oral contraceptives within 30 days prior to first dosing.
26. Use of long-acting estrogen or progestin injections (including progestin-releasing IUDs) or implants within 6 months prior to first dosing.
27. Any other condition that, in the opinion of the investigator, makes the participant unsuitable for study participation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-07-20 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Area under plasma concentration-time curve from time zero to infinity (AUC) for VCT220. | 1 hour pre-dose on D1 and D11, and 0.5h, 1h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 48h, 72h post dose
  Rifampin Cohort
Area under plasma concentration-time curve from time zero to infinity (AUC) for VCT220 | 1 hour pre-dose on D1 and D12, and 0.5h, 1h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 48h, 72h post dose
  Itraconazole Cohort
Maximum observed plasma concentration (Cmax) for VCT220 | 1 hour pre-dose on D1 and D11, and 0.5h, 1h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 48h, 72h post dose
  Rifampin Cohort
Maximum observed plasma concentration (Cmax) for VCT220 | 1 hour pre-dose on D1 and D12, and 0.5h, 1h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 48h, 72h post dose
  Itraconazole Cohort

SECONDARY OUTCOMES:
Number of participants with adverse events | From the 1st dosing day and 1-2 days after last treatment (day 15)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No